CLINICAL TRIAL: NCT01013025
Title: Phave IV, Multicenter, Open-label Study to Collect VANTAS® Implant Retrieval Data From Patients With Advanced Prostate Cancer and Difficult to Remove Implants
Brief Title: Vantas Implant Retrieval Study
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Other Study IDs: 303
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; implant retrieval
MeSH Terms: conditions — Prostatic Neoplasms | interventions — High-Energy Shock Waves; histrelin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with Vantas implant: Patients were enrolled if they had had a Vantas implant placed for treatment of adenocarcinoma of the prostate, and if the patients were scheduled for explant of the implant, and the physician had difficulty locating the implant.
  Interventions: Procedure: Ultrasound or CT or MRI to locate implant

INTERVENTIONS:
Procedure: Ultrasound or CT or MRI to locate implant — Scanning methods (eg, ultrasound, CT, or MRI) were used to locate the implant.
  Other Names: Vantas

SUMMARY:
The main study objective was to collect implant retrieval information in 10 patients using Vantas®, the 50 mg histrelin implant. Patients who had been identified as having a difficult to locate or non-palpable implant were to have been enrolled. Sites were to adhere to the instructions in the Package Insert, which included specialized investigations such as ultrasound, CT, and MRI, to be used for the location and removal of implants.

DETAILED DESCRIPTION:
Up to 50 centers using Vantas, the recently approved histrelin implant as part of their urology practice for treating patients with advanced prostate cancer, were to be identified for participation in this Phase IV post-marketing trial. Up to 10 patients who had been implanted with Vantas at these participating centers, and who had difficult to locate or non-palpable implants at the time of removal, were to be enrolled in this trial. A Screening Visit was to be conducted to consent the patient and to collect basic medical and safety information for patient participation. Upon patient enrollment, up to three subsequent Visits (Visits 1, 2, and 3) were to be conducted (within 2 weeks of the Screening Visit). The investigator was to locate and remove the implant by following the instructions provided in the protocol. Methods for location of the implant included ultrasound, CT, or MRI procedures. The visit at which the implant was successfully located and removed was to be the final study visit for the patient. Upon successful retrieval of the implant or a determination that, per Study Instructions, the implant cannot be located/removed, the study was completed for the patient. No information was to be collected on re-implantation of a new implant. Safety was to be monitored throughout the two week study. Blood samples for testosterone and PSA were only collected at the Screening Visit. The implants removed from the patients were to be returned to Indevus Pharmaceuticals for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Were male patients with adenocarcinoma of the prostate;
* Were age 45 years or older;
* Had received a Vantas® implant;
* Had difficult to locate or non-palpable implant at time of implant retrieval;
* Had the ability to undergo ultrasound, and/or CT, and/or MRI within two weeks of Screening Visit;
* Voluntarily provided Informed Consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

* Major medical or psychiatric illness that would interfere with return visits; patient not suitable (e.g., noncompliance history) for study in opinion of the Investigator or Sponsor;
* Participated in a clinical trial for an investigational agent within 30 days prior to the Screening Visit (unless enrolled in Protocol 301 Extension).

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was planned to include approximately 10 patients with locally advanced or metastatic prostate cancer who satisfied the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The number (and percent) of successfully located and removed implants was the primary outcome measure. | cross-sectional design, data collected at time of explant procedure.